CLINICAL TRIAL: NCT03846518
Title: Comparison of Two Tooth-borne Expanders in Rapid Maxillary Expansion: Dentoalveolar Effects and Impact on Quality of Life
Brief Title: Comparison of Two Tooth-borne Expanders in Rapid Maxillary Expansion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pontifícia Universidade Católica de Minas Gerais (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Principal Investigator, Dauro Douglas Oliveira, Associate professor and program director of Orthodontics, Pontifícia Universidade Católica de Minas Gerais
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: hyraxversusminihyrax
Record Dates: First submitted 2019-02-17; First posted 2019-02-19 (Actual); Last update posted 2020-03-05 (Actual); Status verified 2020-03

CONDITIONS: Malocclusion; Posterior Crossbite
Keywords: palatal expansion technique; adolescent; quality of life
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Intervention Model Description: 2 groups: control group (Hyrax) and experimental group (mini Hyrax)
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hyrax group (Active Comparator): Seventeen patients will be submitted to rapid maxillary expansion (RME) using the Hyrax expander. The activation protocol will be 2 turns a day up to obtain transverse overcorrection.
  Interventions: Device: Hyrax
- mini Hyrax group (Experimental): Seventeen patients will be submitted to rapid maxillary expansion (RME) using the mini Hyrax expander. The activation protocol will be 2 turns a day up to obtain transverse overcorrection.
  Interventions: Device: mini Hyrax

INTERVENTIONS:
Device: Hyrax — Rapid maxillary expansion using the Hyrax expander. Appliance anchorage will be performed by bands adapted to the first maxillary molars and arms of the screw contoured to adapt to palatal faces of the first and second maxillary bicuspids, in wich will be bonded by resin. The screw will be positioned perpendicularly to the palate sagittal midline, between second maxillary bicuspids and first maxillary molars, and 5 mm apically from marginal gingiva of palatal face of the first maxillary molars.The activation protocol will be 2 turns a day up to obtain transverse overcorrection. After the active period of RME, the screws will be fixed with ligature wire and the appliance will be kept as a retainer for 6 months.
  Arms: Hyrax group
Device: mini Hyrax — Rapid maxillary expansion using the mini Hyrax expander. Appliance anchorage will be performed by bands adapted to the first maxillary molars and arms of the screw contoured to adapt to palatal faces of the first and second maxillary bicuspids, in wich will be bonded by resin. The screw will be positioned perpendicularly to the palate sagittal midline, between second maxillary bicuspids and first maxillary molars, and 5 mm apically from marginal gingiva of palatal face of the first maxillary molars. The activation protocol will be 2 turns a day up to obtain transverse overcorrection. After the active period of RME, the screws will be fixed with ligature wire and the appliance will be kept as a retainer for 6 months.
  Arms: mini Hyrax group

SUMMARY:
This study will assess the dentoalveolar effects and impact on quality of life of two types of maxillary expanders in orthodontic patients with permanent dentition, from 12 to 16 years old. Half of participants will be treated using the Hyrax expander, while the other half will use the mini Hyrax expander. The null hypothesis is that there is no difference between dentoalveolar effects and impact on quality of life of the two protocols.

DETAILED DESCRIPTION:
Transverse maxilla deficiency is characterized by narrowing of the maxillary arch with important functional and esthetic impact. In individuals which have not reached bone maturity, a rapid expansion of the maxilla by using tooth-borne expanders as Haas and Hyrax appliance are efficient and safe. A presentation of favorable results for the "mini-Hyrax inverted" expander with a small screw in the transversal correction of the maxilla in patients with cleft lip and palate, besides improving the comfort and the teeth cleaning, provoked an idea of application of this small screw to correct posterior crossbite in individuals without cleft lip and palate. The objective of this study is to compare the dentoalveolar effects and impact on quality of life of two types of maxillary expanders in adolescent patients with permanent dentition and active bone growth. The sample size calculation indicated a total sample of 28 individuals. Taking into account the loss of sample during the study, 34 subjects that have posterior crossbite and age from 12 to 16 years, will be recruited at the Dental School, Pontifical University Catholic of Minas Gerais, Belo Horizonte, Minas Gerais, Brazil. These patients will be randomly divided into two groups, Hyrax and mini Hyrax, with 17 patients each. Digital models of both dental arches will be obtained by intraoral scanning precede the procedure (T0) and at the end of the retention period, after appliance removal (T2). OHIP-14 Oral Health Impact Profile Questionnaires, validated in Portuguese, will be applied before expansion (T0), after an expansion (T1) and at the end of the retention period (T2). In digital dental models, maxillary first and second bicuspids and first molar width, and rotation and inclination of maxillary first bicuspids and first molars will be assessed. After the normality test, the appropriate statistical test will be used in the intergroup comparison. A significance level of 5% will be regarded for all tests.

ELIGIBILITY:
Inclusion Criteria:

* Maxillary permanent dentition, except canines
* Ages ranging from 12 to 16 years old;
* Maxillary constriction associated to posterior crossbite uni or bilateral.

Exclusion Criteria:

* Cleft lip and palate;
* Craniofacial syndromes;
* Carious lesions;
* History of previous orthodontic treatment.

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — Initially the 34 individuals will be separated by sex, thenceforth the randomization to alocation in the groups will be applied. The objetive of it is avoid major difference in sex between the 2 groups.
Enrollment: 34 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-09-18 (Actual); Study Completion 2020-02-27 (Actual)

PRIMARY OUTCOMES:
Maxillary first molars width. Scale in millimeters and one decimal place. | 6 months
  Distance between centroid points of maxillary first molars
Maxillary first bicuspid width. Scale in millimeters and one decimal place. | 6 months
  Distance between centroid points of maxillary first bicuspids
Maxillary second bicuspid width. Scale in millimeters and one decimal place. | 6 months
  Distance between centroid points of maxillary second bicuspids
Maxillary first molas angulation. Scale in degrees and one decimal place. | 6 months
  Angulation formed, in occlusal view, by intersection of the lines resulted of the link between mesial-buccal cuspid tip and mesial-palatal cuspid tip of each molar.
Maxillary first bicuspids angulation. Scale in degrees and one decimal place. | 6 months
  Angulation formed, in occlusal view, by intersection of the lines resulted of the link between buccal cuspid tip and palatal cuspid tip of each bicuspid
Maxillary first molas inclination. Scale in degrees and one decimal place. | 6 months
  Angulation formed, in coronal view, by intersection of the lines resulted of the link between mesial-buccal cuspid tip and mesial-palatal cuspid tip of each molar
Maxillary first bicuspids inclination. Scale in degrees and one decimal place. | 6 months
  Angulation formed, in coronal view, by intersection of the lines resulted of the link between buccal cuspid tip and palatal cuspid tip of each bicuspid

SECONDARY OUTCOMES:
Quality of life evaluation using questionnaires | 2 weeks (2 times: 0 and 2 weeks after insert of device) and 6 months (after removal of device)
  Oral Health Impact Profile (OHIP-14) will be used to evaluate the quality of life of the patients before, during and after treatment. Fourteen items that explore seven dimensions of impact: functional limitation, physical pain, psychological discomfort, physical disability, psychological disability, social disability and handicap. The responses will be classified using the Likert scale with five options ranging from "never" (0) to "very often" (4). Higher values represent higher levels of impact on each dimension.
Discomfort evaluation using questionnaires | 24 hours (4 times: 0, 24, 48 and 72 hours after insert of device) and 1 week (2 times: 1 and 2 weeks after insert of device)
  A Visual Analog Scale will be used from 0 to 100. Scale in millimeters and one decimal place. Higher values represent higher level of pain. The 0 point represents absence of pain and the 100 point represents the maximum pain that patient imagines is possible exist.

CONTACTS AND LOCATIONS:
Overall Officials: Dauro D Oliveira, PhD, Study Chair — Associate professor and program director of Orthodontics
Locations (1):
- Pontifícia Universidade Católica de Minas Gerais, Belo Horizonte, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No